CLINICAL TRIAL: NCT05362097
Title: Analysis of the Reliability and Validity of the Chinese Version of Child Cough-specific Quality of Life Questionnaire(CC-QoL)
Brief Title: Analysis of the Reliability and Validity of the Chinese Version of CC-QoL
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD-LSUN3
Record Dates: First submitted 2022-04-15; First posted 2022-05-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Chronic Cough
Keywords: reliability validity Cc-QOL
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The reliability and validity of the Chinese version of CC-QoL — Cc-qol, LCQ, and VCD were repeated 1-2 times before and 1-13 weeks after treatment.

SUMMARY:
At present, there is no research scale designed for the quality of life of children with chronic cough in China, most of them use the cough scale designed for adults to evaluate the quality of life of children. In China, more and more attention has been paid to evaluate and improve the quality of life of children with chronic cough, but cough specific quality of life measurement tools for adults and parents are mostly used, and the Chinese translation version of CQLQ and LCQ is still the main method. There is still no cough specific quality of life measurement tool for children with chronic cough in China. Cc-qol, a specific scale for chronic cough in children, has not been promoted, and no relevant verification of the applicability, validity and reliability of the Chinese version has been found. Therefore, this study aims to verify and compare the applicability, reliability and validity of CC-QOL Chinese version in China through questionnaire survey and follow-up of children with chronic cough.

DETAILED DESCRIPTION:
Descriptive Score: CC-QOL, CET,VAS, Peds-QOL,SCAS and Verbal category Score (VCD); descriptive score: DESCRIPTIVE score; descriptive score: DESCRIPTIVE score; descriptive score: DESCRIPTIVE score; To evaluate the reliability and validity of Cc-QOL in evaluating children's quality of life in China, Compare and analyze Leicester cough questionnaire(LCQ) and child chronic cough-specific quality of life measure Cc-qol was used to evaluate the quality of life in children with chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 7-14；
* 2.Disease duration > 4 weeks；
* 3.Spontaneous cough as the main or only clinical symptom。

Exclusion Criteria:

* Chest X-ray was unremarkable, excluding cystic fibrosis, typical asthma or dyspnea, and other underlying diseases.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The childr who conforms to the definition of "Chronic cough in children in the Guidelines for the Diagnosis and Treatment of Chronic Cough in Chinese Children (Revised in 2013)".
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-03-05 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Validity | At first visit, before medication, 2 weeks and 6 weeks after treatment initiation
  Validity mainly evaluates the accuracy, validity and correctness of the scale, that is, the deviation between the measured value and the true target value.Validity is meant to reflect whether a measuring tool can effectively measure what it is intended to measure, that is, the extent to which the actual measured results agree with the expected results.
Reliability | At first visit, before medication, 2 weeks and 6 weeks after treatment initiation
  Reliability refers to the reliability, stability and consistency of the survey results, that is, accuracy.It is generally believed that reliability reflects the variation degree caused by measurement error or observation error, that is, random error.Common indicators:
  Common indicators:
  It is generally believed that Cronbach's alpha should be above 0.7. Retest reliability: the same questionnaire is used to measure the same group of respondents repeatedly at different times, and the consistency between the two results is retest reliability.

SECONDARY OUTCOMES:
Sensitivity | At first visit, before medication, 2 weeks and 6 weeks after treatment initiation
  To evaluate the sensitivity of the questionnaire to measurements before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China